CLINICAL TRIAL: NCT06048965
Title: An Expert Panel Consensus Statement on the Management of Menopause in the Asia-Pacific Using Modified Delphi Methodology
Brief Title: Asia Pacific Menopause Federation Menopause Consensus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: APMFMenopause2023
Record Dates: First submitted 2023-08-29; First posted 2023-09-21 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Menopause; Menopause Related Conditions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Expert group
  Interventions: Other: No intervention to be performed

INTERVENTIONS:
Other: No intervention to be performed — No intervention to be performed. Anonymous survey only.

SUMMARY:
The aim of this study is to achieve expert consensus on the management of menopause in the Asia-Pacific

DETAILED DESCRIPTION:
The aim of this study is to achieve expert consensus on the management of menopause in the Asia-Pacific. The experience of the menopause is deeply rooted in sociocultural perceptions unique to each population. Thus, the management of menopausal symptoms and other conditions related to the menopause also vary from region to region.

The investigators will use a modified Delphi method involving the participation of experts from various countries in the Asia-Pacific. The objective of this study is to achieve consensus on various aspects of the management of the menopause in the Asia-Pacific.

This study will involve several rounds of Delphi surveys, administered via Google Forms, Microsoft Word or PDF. Each survey questionnaire contains

1. Questions on basic demographic information
2. Statements on areas of concern in the management of the menopause; each participants vote on to what extent they agree or disagree with the statement on a Likert scale.
3. Questions on the participants' usual clinical practice in treating menopause Multiple survey rounds will be held until agreement on the statements and stability is achieved.

ELIGIBILITY:
Inclusion Criteria:

Experience in treating menopause

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physicians with experience in treating menopause
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-20 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who vote for the same option on a series of survey questions | 2023-2024

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No